CLINICAL TRIAL: NCT03339440
Title: A Randomized Trial of an Integrated Clinic-community Intervention in Children and Adolescents With Obesity
Brief Title: A Trial of an Integrated Clinic-community Intervention in Children and Adolescents With Obesity (Hearts and Parks)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00086684
Record Dates: First submitted 2017-10-30; First posted 2017-11-13 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Childhood Obesity; Pediatric Obesity; Quality of Life; Cardiovascular Risk Factor
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: The investigators will use a two-arm, randomized crossover controlled trial to compare routine primary care management of childhood obesity versus a novel clinic/family/community partnership program to treat childhood obesity. This design will allow for a randomized comparison of Group 1 (6-month standard control) to Group 2 (immediate 6-month intervention program) and to Group 3 (delayed crossover intervention on the standard control group). The design will also allow the investigators to observe intervention effects at 3 months in both intervention groups (Groups 2 and 3), and to track Group 2 for 6 additional months after active intervention to assess whether health benefits seen at 6 months were sustained to 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients in this group will be receiving the Hearts and Parks intervention.
  Interventions: Behavioral: Hearts & Parks
- Control Group (No Intervention): Patients in this group will continue receiving standard of care.

INTERVENTIONS:
Behavioral: Hearts & Parks — The Hearts & Parks intervention will be looking to evaluate how different types of physical activity and nutrition education and support (in addition to normal clinical care) through attendance and participation in the Duke Healthy Lifestyles/Bull City Fit clinic/community program, affect children's health. The investigators will be looking at changes in BMI, physical activity, nutrition and overall health.
  Arms: Intervention Group

SUMMARY:
The investigators propose a randomized controlled effectiveness trial to evaluate the integrated clinic-community model of child obesity treatment as compared with routine primary care.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate how different types of physical activity and nutrition education and support (in addition to normal clinical care) affect children's health. The investigators will be looking at changes in child BMI, physical activity, nutrition, and overall health. The investigators also hope to better understand biological differences in metabolism and the microbiome (the bacteria that grows normally on and in the body) in children with high BMI who are making lifestyle changes.

ELIGIBILITY:
Inclusion Criteria:

* Child age 5-18 years
* Child body mass index ≥ 95th %ile
* Parent can speak and read in English or Spanish
* Parent ownership of a device that is able to receive and send text messages

Exclusion Criteria:

* Live farther than a 20-mile radius from the Healthy and Fit program site
* Endogenous or genetic cause of obesity
* Taking a medication that causes weight gain
* Participation in a pediatric weight management program within 12 months
* Parent or child significant health problem that would limit participation
* Enrollment is above the max weekly enrollment of 60 participants/week)
* Reported or planned pregnancy

Opt-out Criteria

• Primary care physician opts patient out of study for reasons including: severe obesity, urgent co-morbidities, parental unwillingness to be contacted by a research assistant, or at physician clinical judgment.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 327 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in z-BMI | Baseline, 6 months
Change in heart rate | baseline, 12 months
Number of subjects enrolled versus number of subjects who meet min. participation criteria | 12 months
  As measured by enrollment logs
Change in molecular pathways dysregulated in pediatric obesity | Baseline, 6 months
  Stool and blood samples
Physical activity | Up to 12 months
  child physical activity; objectively tracked with fitness tracker
Change in child fitness | baseline, 3 months, 12 months
  3 minute bench stepping test
Change in Child Quality of Life | baseline, 3 months, 12 months
  Composite score of Sizing Me Up Questionnaires
Change in Body Appreciation | baseline, 3 months, 12 months
  Body appreciation scale 13-item questionnaire (1. Never, 2. Seldom, 3. Sometimes, 4. Often, 5. Always)
Change in FLASHE Food and Activity Screener Scores | Baseline, 6 months, 12 months
  Questionnaire about child and parent nutrition and activity habits
Change in fasting lipid profile | Baseline, 6 months, 12 months
Change in fasting glucose | Baseline, 6 months, 12 months
Change in alanine aminotransferase (A1) | Baseline, 6 months, 12 months
Change in child quality of life (2) | baseline, 3 months, 12 months
  PROMIS Questionnaire (not composite score)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Armstrong, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Duke Children's Primary Care Roxboro Street, Durham, North Carolina
  - Durham Pediatrics at North Duke Street, Durham, North Carolina
  - Regional Pediatrics - North Durham, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh K, Armstrong SC, Wagner BE, Counts J, Skinner A, Kay M, Li JS, Shah S, Zucker N, Neshteruk C, Story M, Suarez L, Kraus WE, Zizzi AR, Dunn J. Physical activity and sleep changes among children during the COVID-19 pandemic. NPJ Digit Med. 2024 Mar 16;7(1):70. doi: 10.1038/s41746-024-01041-8. PMID 38493216
- [Derived] Dunn J, Singh K, Armstrong S, Wagner B, Counts J, Skinner A, Kay M, Li J, Shah S, Zucker N, Neshteruk C, Suarez L, Kraus W, Zizzi A. Physical activity and sleep changes among children with obesity during a period of school closures related to the COVID-19 pandemic. Res Sq [Preprint]. 2023 Sep 13:rs.3.rs-3293474. doi: 10.21203/rs.3.rs-3293474/v1. PMID 37790374
- [Derived] Neshteruk CD, Zizzi A, Suarez L, Erickson E, Kraus WE, Li JS, Skinner AC, Story M, Zucker N, Armstrong SC. Weight-Related Behaviors of Children with Obesity during the COVID-19 Pandemic. Child Obes. 2021 Sep;17(6):371-378. doi: 10.1089/chi.2021.0038. Epub 2021 Apr 26. PMID 33902326
- [Derived] Armstrong SC, Windom M, Bihlmeyer NA, Li JS, Shah SH, Story M, Zucker N, Kraus WE, Pagidipati N, Peterson E, Wong C, Wiedemeier M, Sibley L, Berchuck SI, Merrill P, Zizzi A, Sarria C, Dressman HK, Rawls JF, Skinner AC. Rationale and design of "Hearts & Parks": study protocol for a pragmatic randomized clinical trial of an integrated clinic-community intervention to treat pediatric obesity. BMC Pediatr. 2020 Jun 26;20(1):308. doi: 10.1186/s12887-020-02190-x. PMID 32590958